CLINICAL TRIAL: NCT02930993
Title: A Safety and Efficacy Study of Autologous T Cells Engineered to Express Chimeric Antigen Receptor Targeting Mesothelin in Patients With Recurred or Metastatic Malignant Tumors
Brief Title: Anti-mesothelin CAR T Cells for Patients With Recurrent or Metastatic Malignant Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Meitan General Hospital (Other)
Collaborators: Marino Biotechnology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jinwen Sun, director of Department of General Surgery and Surgical Oncology, China Meitan General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K16-4
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Mesothelin Positive Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- anti-mesothelin CAR T cells (Experimental): Dose escalation study aimed to assess the safety and efficacy of anti-mesothelin CAR T cells.
  CAR T dosage ranging from 5×10^4 /kg to 1×10^7 /kg will be tested .
  Interventions: Biological: anti-mesothelin CAR T cells

INTERVENTIONS:
Biological: anti-mesothelin CAR T cells — Patients will be received a three-day regimen of chemotherapy consisting of cyclophosphamide aimed to deplete the lymphocytes. 1 to 4 days after lymphodepletion, patients are intravenously infused with anti-mesothelin CAR T cells in a three-day split-dose regimen (day0,10%; day1, 30%; day2, 60%).

SUMMARY:
This is a single-arm, open-label, one center, dose escalation clinical study, to determine the safety and efficacy of infusion of autologous T cells engineered to express chimeric antigen receptor targeting mesothelin in adult patients with mesothelin positive, recurrent or metastatic malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

1. patients with mesothelin positive, recurrent or metastatic malignant tumors , including but not limited to pancreatic adenocarcinoma, ovarian cancer, or pleural mesothelioma.
2. relapsed or metastatic after standard treatment
3. measurable tumors by RECIST1.1 standard
4. patients are 18 to 70 years old.
5. life expectancy > 3months.
6. KPS ≥70.
7. satisfactory major organ functions: adequate heart function with LVEF≥50%; no obvious abnormities in ECG; pulse oximetry ≥ 90%; cockcroft-gault creatinine clearance≥40 ml/min; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3ULN; Bilirubin ≤2.0 mg/dl .
8. Blood: Hgb ≥ 80 g/L, ANC ≥ 1×10^9/L, PLT ≥ 50×10^9/L.
9. women of reproductive potential must have a negative pregnancy test. Male and female of reproductive potential must agree to use birth control during the study and one year post study.

Exclusion Criteria:

1. patients with a prior history of autoimmune disease or other diseases who need long-term use of systemic hormone drug or immunosuppressive therapy
2. active infection.
3. HIV positive.
4. active hepatitis B virus infection or hepatitis C virus infection.
5. currently enrolled in other study.
6. patients, in the opinion of investigators, may not be eligible or are not able to comply with the study.
7. patients who have allergic disease, or are allergic to T cell products or other biological agents used in the study.
8. patients whose tumors have metastasized to bone marrow, or have clinical signs of bone metastasis, such as bone and joint pain .
9. patients who have brain metastasis or signs of brain metastasis, such as loss of self-consciousness.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
safety of infusion of autologous anti-mesothelin CAR T cells as assessed by the incidents of treatment related adverse events per NCI CTCAE V4.0 | 2 years
  incidents of treatment related adverse events per NCI CTCAE V4.0

SECONDARY OUTCOMES:
treatment response rate of anti-mesothelin CAR T cells | 4 weeks
  Defined as the overall response rate (ORR), the proportion of patients who achieved complete remission (CR), partial remission (PR), stable disease (SD), or progressive disease (PD) based on the response evaluation criteria in solid tumor version 1.1 (RECIST1.1).
progression free survival | 6 months
overall survival | 2 years
proliferation of anti-mesothelin CAR T cells in patients | 6 months
  measured by quantitative PCR and flow cytometry
activation of anti-mesothelin CAR T cells in patients | 6 months
  measured by blood cytokine levels after CAR T cell infusion
persistence of anti-mesothelin CAR T cells in patients | 1 year
  measured by quantitative PCR and flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Jinwen Sun, MD, Principal Investigator — China Meitan General Hospital
Locations (1):
- China Meitan General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided